CLINICAL TRIAL: NCT05163119
Title: Randomized Trial on Mobile Technology and Young Drivers' Cellphone Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Motao Zhu (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Ohio State University (Other); University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Motao Zhu, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001601; R01HD102439 (NIH)
Record Dates: First submitted 2021-12-05; First posted 2021-12-20 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cell Phone Use; Automobile Driving
Keywords: Texting; Driving; Mobile Technology
MeSH Terms: conditions — Cell Phone Use | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): Commercial cell-phone blocking app installed on smartphone, but app will be inactive.
- Commercial Cellphone-Blocking App (Experimental): Commercial cellphone-blocking app that blocks handheld cellphone use while driving, but allows emergency calls and phone use after pressing the passenger button will be installed on smartphone.
  Interventions: Behavioral: Commercial Cellphone-Blocking App (Active)
- Driving Mode (Experimental): Driving mode blocks handheld phone use while driving or facilitates hands free use (exact functionality dependent on smartphone type and service provider).This group will also have the commercial cell-phone blocking app installed on smartphone, but app will be inactive.
  Interventions: Behavioral: Driving Mode

INTERVENTIONS:
Behavioral: Commercial Cellphone-Blocking App (Active) — The Fleetsafer app, which is a commercial cellphone app that uses a cellphone's standard sensors and function to block handheld cellphone use while driving, will be downloaded on the participant's smartphone.
  Arms: Commercial Cellphone-Blocking App
Behavioral: Driving Mode — Apple's "Do Not Disturb" driving mode provided by Apple for iPhones or Google Do Not Disturb, Verizon Messages +, Android Auto or have another app, called LifeSaver installed on their Android phone (collectively referred to as driving modes; the specific driving mode for participants in this arm will be determined based on smartphone type and service provider).
  Arms: Driving Mode

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial to determine the effects of a cellphone app and a driving mode intervention on driving behavior in drivers aged 18-24 years.

DETAILED DESCRIPTION:
For this study, 1200 teens aged 18-24 years will be randomized into one of three study groups for 6 months. Researchers aim to evaluate the effectiveness of commercial cellphone-blocking apps and driving mode interventions on cellphone use while driving and evaluate the effectiveness of commercial cellphone-blocking apps and driving mode interventions on high-risk driving events.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-24 years of age at time of recruitment
* Must have ownership and exclusive access to a passenger vehicle
* Must have car insurance with at least state-minimum coverage
* Must live in Greater Columbus (Ohio) area
* Must drive at least 2 days a week on average
* Must have functioning iPhone or Android smartphone with an active phone service account (Ex: Verizon, AT&T, etc.)
* Must self-report handheld calling or texting while driving (≥ 1 time/week)
* Must not be enrolled in another driving-related research study during the study period.
* Must be willing to be randomized and comply with study requirements
* Must have no plans to change cellphones or vehicles in next 6 months or agree to transfer FleetSafer app/DriveCam if they change cellphones or vehicles
* Must speak and read English

Exclusion Criteria:

* Drivers under 18 years of age
* Drivers holding learner's permits
* Drivers who share a vehicle with a family member or others
* Infrequent drivers (Drive 2 days a week or less)
* Participants from the pilot R21 project
* Current users of a cellphone-blocking app or driving mode who do not agree to uninstall/de-activate the app for the duration of participation in the study
* Current users of a car insurance monitoring device (physical device or app)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Calling, texting, and handheld cell phone use while driving | 5-month intervention period
  Number of calling occurrences, texting occurrences, and handheld phone use occurrences, per 1,000 miles driven. Higher numbers signify more calling, texting, and handheld cell phone use.
High-risk driving events | 5-month intervention period
  Total number of high-risk driving events (e.g., hard-braking, sudden acceleration, swerving) per 1,000 miles driven. Higher numbers signify more high-risk driving events.

CONTACTS AND LOCATIONS:
Overall Officials: Motao Zhu, Principal Investigator — Abigail Wexner Research Institute at Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No